CLINICAL TRIAL: NCT05931939
Title: Ileal Interposition to the Treatment of Weight Regain After Roux-en-Y Gastric Bypass: a Randomized Controlled Trial
Brief Title: Laparoscopic Ileal Interposition and Weight Regain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer-Aguiar, MD, Principal Investigator, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ileal interposition
Record Dates: First submitted 2023-05-07; First posted 2023-07-06 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized intervention study, comparing the effect of revisional surgery by laparoscopic Ileal Interposition with traditional surgical technique
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ileal Interposition (Experimental): Interposition ileal surgery group Procedure/Surgery: Bariatric surgery
  Interventions: Procedure: Ileal Interposition
- Traditional surgical technique (Active Comparator): Conventional revisional surgery group Procedure/Surgery: Bariatric surgery
  Interventions: Procedure: Traditional surgical technique

INTERVENTIONS:
Procedure: Ileal Interposition — Bariatric surgery by laparoscopic Ileal Interposition
  Arms: Ileal Interposition
Procedure: Traditional surgical technique — Bariatric surgery by laparoscopic traditional technique
  Arms: Traditional surgical technique

SUMMARY:
The investigators will study the Ileal interposition to the treatment of weight regain after Roux-en-Y gastric bypass, assessing weight loss, body composition, quality of life, metabolic biomarkers, inflammatory biomarkers, and incretin hormones

DETAILED DESCRIPTION:
This prospective, controlled, randomized intervention study will investigate the Ileal interposition to the treatment of weight regain after Roux-en-Y gastric bypass, assessing weight loss, body composition, health-related quality of life, metabolic biomarkers, inflammatory biomarkers, and incretin hormones. The participants will also be assessed for alcohol abuse, depressive symptoms, level of physical activity, eating disorder symptoms, and dumping syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to initial laparoscopic after initial Roux-en-Y gastric bypass for at least 3 years
* Loss of excess weight between 60 to 80%
* Rate of weight regain ≥60%
* Body mass index ≥ 40 kg/m2 or ≥ 35 kg/m2, with at least 2 comorbidities associated with obesity
* Present a previous evaluation by the multidisciplinary team with a favorable opinion of the revision surgery.

Exclusion Criteria:

* Active chemical dependency on alcohol and/or illicit drugs
* Severe psychotic or depressive disorder or history of suicide attempts in the last 12 months
* Eating behavior disorder (uncontrolled)
* Secondary causes of obesity
* Pregnancy
* Severe organ failure
* Active neoplastic
* Infectious or inflammatory disease
* Severe coagulopathy
* High anesthetic-surgical risk
* Intellectual inability
* Lack of preoperative follow-up

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes of weight loss of participants after Ileal interposition surgery as measured by weight in kilograms | Change from baseline and after 6 months post-surgery
  Weight loss will be obtained as the difference between preoperative weight and minimum postoperative weight in kilograms
Changes of Health-related quality of life of participants after Ileal interposition surgery as reported by 36-Item Short-Form Health Survey questionnaire | Change from Baseline and after 6 months post-surgery
  Health-related quality of life will be assessed using the 36-Item Short-Form Health Survey questionnaire

SECONDARY OUTCOMES:
Changes of weight loss of participants after Ileal interposition surgery as measured by weight in kilograms | Change from baseline and after 3, 6, and 12 months post-surgery
  Weight loss will be obtained as the difference between preoperative weight and minimum
Change of body composition of participants after Ileal interposition surgery as measured by lean and fat mass in kilograms | Change from baseline and after 6 and 12 months post-surgery
  Body composition will be assessed through dual X-ray absorptiometry (DXA)
Change of metabolic profile of participants after Ileal interposition surgery as assessed by serum levels of glucose and insulin | Change from baseline and after 6 and 12 months post-surgery
  Blood sample collection will include serum levels of glucose and insulin
Change of inflammatory biomarkers and incretin hormones of participants after Ileal interposition surgery as assessed by serum levels of tumor necrosis factor-alpha, interleukin-6, ghrelin, and glucagon-like peptide-1. | Change from baseline and after 6 months post-surgery
  Blood sample collection will include serum levels of tumor necrosis factor-alpha, interleukin-6, ghrelin, and glucagon-like peptide-1.
Changes in alcohol abuse of participants after Ileal interposition surgery as reported by Alcohol Use Disorders Identification Test | Change from baseline and after 6 and 12 months post-surgery
  Alcohol abuse will be assessed using the Alcohol Use Disorders Identification Test
Changes in depressive symptoms of participants after Ileal interposition surgery as reported by Beck Depression Inventory | Change from baseline and after 6 and 12 months post-surgery
  Depressive symptoms will be assessed using the Beck Depression Inventory questionnaire
Changes in the level of physical activity of participants after Ileal interposition surgery as reported by the International Physical Activity Questionnaire | Change from baseline and after 6 and 12 months post-surgery
  Levels of physical activity will be assessed using the International Physical Activity Questionnaire
Changes in the eating disorder symptoms of participants after Ileal interposition surgery as reported by the Eating Disorder Examination Questionnaire | Change from baseline and after 6 and 12 months post-surgery
  Eating disorder symptoms will be assessed using the Eating Disorder Examination Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Guilherme Kraemer-Aguiar, PhD, Principal Investigator — State University of Rio de Janeiro; Paulo Roberto G Falcão Leal, MD, Principal Investigator — State University of Rio de Janeiro; Karynne G Grutter Lopes, PhD, Principal Investigator — State University of Rio de Janeiro
Locations (1):
- State University of Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No